CLINICAL TRIAL: NCT03531606
Title: The Effects of Mechnikov Probiotics on Symptom and Surgical Outcome After Anterior Resection of Colon Cancer; Double-blind, Randomized, Placebo-controlled Trial
Brief Title: The Effects of Mechnikov Probiotics on Symptom and Surgical Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kye Bong-Hyeon (Other)
Responsible Party: Sponsor-Investigator, Kye Bong-Hyeon, Associate Professor, The Catholic University of Korea
Organization: The Catholic University of Korea (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY_Mpro3
Record Dates: First submitted 2018-04-15; First posted 2018-05-22 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Sigmoid Colon Cancer
MeSH Terms: conditions — Sigmoid Neoplasms

STUDY DESIGN:
Intervention Model Description: This study has been designed for randomized, double Blinded, placebo clinical trial.
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Using placebo comparator with experimental one, it will be compared between two group for comparison of placebo comparator with experimental one.
  The patients enrolled into expeimental group will take one pack of 'Mechnicov probiotics' twice a day for 4 weeks from 1 week before surgery.
  (1 week before surgery and 3 weeks after surgery)
  The patients in placebo and experimental group should take a part in this clinical trial under the condition of 'anterior resection of colon cancer'
  Interventions: Drug: Mechnicov probiotics
- Placebo comparator (Placebo Comparator): Using placebo comparator with experimental one, it will be compared between two group for comparison of placebo comparator with experimental one.
  The patients enrolled into placebo comparator group will take one pack of 'Placebo' which is composed of lactose and simulates a 'Mechnicov probiotics' twice a day for 4 weeks from 1 week before surgery.
  (1 week before surgery and 3 weeks after surgery)
  The patients in placebo and experimental group should take a part in this clinical trial under the condition of 'anterior resection of colon cancer'
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mechnicov probiotics — Using placebo comparator with experimental one, it will be compared between two group for comparison of placebo comparator with experimental one.
  The patients enrolled into expeimental group will take one pack of 'Mechnicov probiotics' twice a day for 4 weeks from 1 week before surgery.
  (1 week before surgery and 3 weeks after surgery)
  The patients in placebo and experimental group should take a part in this clinical trial under the condition of 'anterior resection of colon cancer'
  Other Names: Anterior resection
  Arms: Experimental
Drug: Placebo — Using placebo comparator with experimental one, it will be compared between two group for comparison of placebo comparator with experimental one.
  The patients enrolled into expeimental group will take one pack of 'Mechnicov probiotics' twice a day for 4 weeks from 1 week before surgery.
  (1 week before surgery and 3 weeks after surgery)
  The patients in placebo and experimental group should take a part in this clinical trial under the condition of 'anterior resection of colon cancer'
  Other Names: Anterior resection
  Arms: Placebo comparator

SUMMARY:
The purpose of this clinical trial study was to evaluate the prevalence of colon cancer among the symptom (s) of anterior resection syndrome that may occur after surgery in patients for efficacy and safety in Metchnik probiotic ingestion.

DETAILED DESCRIPTION:
The purpose of the clinical trial is to evaluate the efficacy and safety of the syndrome that may occur after colon cancer surgery, To evaluate the efficacy and safety of the improvement effect of the defecatory activity on the improvement of the Medienkov probiotics biotics on the patients who have the deficit function and planned to surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female aged 20 to over 75 years old
2. As histologically and radiologically diagnosed S colon cancer, those who is scheduled for anterior resection
3. Those who have been agreed to participate in this trial (through Informed consent) before initiation of clinical trial.

Exclusion Criteria:

1. Those who have metastatic colorectal cancer screening
2. Those who have urinary incontinence or fecal incontinence
3. Those who received preoperative chemotherapy or radiotherapy
4. Those who have a history of severe cerebral vascular disease (cerebral infarction, cerebral hemorrhage, etc.), severe cardiac disease (unstable angina pectoris, myocardial infarction, arrhythmia requiring heart failure heart failure therapy)
5. Those who have neurologist or psychologically important psychiatric history or current disease
6. Those who have alcohol addiction, substance abuse
7. Those who have Immune system, infectious infectious disease, gastrointestinal tract disease patients (inflammatory bowel disease)
8. Those who have uncontrolled hypertension, diabetes patients
9. Those who have creatinine with more than twice from normal upper limit in site
10. Those who have AST(GOT) or ALT(GPT) with more than three times from normal upper limit in site
11. Those who have probiotics, antibiotics, continually within the last one week
12. Those who is pregnant women, breastfeeding women and have pregnancy plans or do not agree to appropriate contraception methods choice
13. Those who have been participated within three months or have plans to participate in another clinical trial after the start of this clinical trial
14. under the investigator's judgment, those who is not qualified to participate this clinical trial

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2016-12-12 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Anterior resection syndrome improvement change | 1 week before surgery, 4 weeks after surgery, 5 weeks after surgery
  3 times performed through questionnaire

SECONDARY OUTCOMES:
Bowel examination | 4 weeks after surgery, 5 weeks after surgery
  2 times performed through questionnaire
Quality of Life of Cancer Patients(EORTC QLQ-C30) | 1 week before surgery, 4 weeks after surgery
  2 times performed through questionnaire
Markers related Inflammation | 1 week before surgery, 4 weeks after surgery
  WBC, Neutrophil, lymphocyce, monocyte, Plt count, neutrophil-lymphocyte ratio
NSI(Nutritional Screening Index) | 1 week before surgery, 1.5 weeks after surgery, 4 weeks after surgery
  PG-SGA: Patient-Generated Subjective Global Assessment
Clavien-Dindo Classification | 1 week after surgery, 1.5 weeks after surgery, 4 weeks after surgery
  Assessment through "Clavien-Dindo Classification"
NGS, SCFA | 1 week before surgery, 1 week after surgery, 4 weeks after surgery, 5 weeks after surgery
  NGS(New Generation Sequencing), SCFA(Short-Chain Fatty Acid)
Other biomarkers | 1 week before surgery, 4 weeks after surgery
  Zonulin, other Cytokines

CONTACTS AND LOCATIONS:
Overall Officials: SungSik Jang, Ph.D, Study Director — R &D
Locations (1):
- In Kyu Lee, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No